CLINICAL TRIAL: NCT01651585
Title: In Utero Treatment of Cytomegalovirus congénitale Infection With Valacyclovir : Prospective Multicenter Nonrandomized Trial
Brief Title: In Utero Treatment of Cytomegalovirus congénitale Infection With Valacyclovir
Acronym: CYMEVAL2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P070708
Record Dates: First submitted 2012-07-25; First posted 2012-07-27 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Foetuses Infection; Cytomegalovirus (CMV)Infection
Keywords: viral disease; cytomegalovirus infection; is the first cause; of congenital; neurological handicap; of infectious origin.
MeSH Terms: conditions — Cytomegalovirus Infections; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Valacyclovir arrow (Experimental): Experimental : Valacyclovir arrow 500mg give Valacyclovir arrow to all participants (open phase)
  Interventions: Drug: Valacyclovir arrow

INTERVENTIONS:
Drug: Valacyclovir arrow — dosage form:500mg, dosage:8g/day, frequency: 4 a day duration: 23 weeks maximum

SUMMARY:
The infection with cytomegalovirus (CMV) is the first cause of congenital neurological handicap of infectious origin. It is probable that the néonatale viral load is correlated with becoming of infected new-born babies. Among the active antiviral treatments against CMV, valacyclovir is the only whose fœtal and maternal tolerance was evaluated during the pregnancy. Its harmlessness and its aptitude to decrease the CMV viral load justify to evaluate it in a study. Decrease the fœtal viral load could make possible to decrease symptomatology néonatale in a group of infected fœtuses.

DETAILED DESCRIPTION:
The infection with cytomegalovirus (CMV) is the first cause of congenital neurological handicap of infectious origin. It is probable that the néonatale viral load is correlated with becoming of infected new-born babies. Among the active antiviral treatments against CMV, valacyclovir is the only whose fœtal and maternal tolerance was evaluated during the pregnancy. Its harmlessness and its aptitude to decrease the CMV viral load justify to evaluate it in a study. Decrease the fœtal viral load could make possible to decrease symptomatology néonatale in infected fœtuses.

To evaluate the effect of a treatment by valacyclovir injected per bone to the mother in the cases of proven fœtal infection with CMV (positive PCR CMV in the amniotic liquid) and presenting cerebral extra echographic signs being able to be allotted to the infection.

The main objective is to observe a reduction in the number of unfavourable exits (symptomatic children at birth) and a reduction in the number of medical interruptions of pregnancy practised for fœtal anomalies.

The secondary objective is a reduction of the CMV viral load in the blood of the cord taken at birth.

The patients included will be treated. The observance will be evaluated. Taking into consideration our preliminary study, a difference of 20% between the 2 groups can be discounted. The number calculated of subjects to include in the test in order to guarantee a power of 80% to him is of 43. Recruitment will be carried out in a multicentric way. The necessary duration of inclusion will be 36 months

The comparison of the two treatments will be carried out on the composite principal criterion according to : proportion of pregnancies with unfavourable exit (symptomatic children at birth or medical interruptions of pregnancy practised for which has appeared cerebral echographic anomalies in connection with the fœtal infection with CMV).

The secondary criteria of judgement will be : the viral load in the blood of the cord of the newborns infected in utero by CMV, the compliance and the criteria of tolerance.

ELIGIBILITY:
Inclusion criteria :

* Age ≥ 18 years,
* Fœtal Infection with CMV authenticated by the positivity of the research of the viral genome by PCR in the amniotic liquid,
* Echographic Assessment revealing at least one cerebral extra anomaly being able to be in connection with the infection with CMV,
* And/or one isolated cerebral anomaly :

  * Ventriculomégalie measured with the ventricular crossroads < 15mm
  * Signs of lenticulo-striated vasculopathy
  * Intraparenchymateuses calcifications
  * Intra-ventricular adherences
* And/or biological signs of generilazed infection to CMV :

  * fetal viremia > 3000 copies/ml
  * platelet < 100 000/cc
* Absence of request for termination of pregnancy from the start,
* Acceptance of a strict follow-up by a Multi-field Center of Prenatal diagnosis and of an optimal observance of the founded treatment,
* Collection of the written assent to take part in the test.
* Affiliation with a mode of social security or equivalent.

Exclusion criteria :

* Not affiliation with a mode of social security (profit or having right)
* Patient of less than 18 years,
* Patient presenting another pathology obstetrical or medical (in particular hepatic or renal) preexistent to tracking or contra-indicating the use of valacyclovir,
* Patientes whose fœtus does not present any echographic sign being able to be in connection with the infection with CMV,
* Patientes whose fœtus presents at least one cerebral echographic anomaly :

Ventriculomégalie measured with the ventricular crossroads ≥ 15mm Hyperechogenicity periventriculaire Hydrocephaly Microcephaly Increase cuts large retro-cérébelleuse cistern Hypoplasy vermienne Porencephaly Lissencephaly Cysts périventriculaires Hypoplasy of the callous body

* Patient under any other active antiviral treatment against CMV,
* Patient taking part in another therapeutic test,
* Patient refusing to sign the enlightened assent,
* Patient formulating a request for medical interruption of pregnancy before inclusion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-07; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
pregnancies with unfavourable exit | 24 hours
  pregnancies with unfavourable exit (symptomatic children at birth or medical interruptions of pregnancy practised for which has appeared cerebral echographic anomalies in connection with the fœtal infection with CMV) at 24 hours

SECONDARY OUTCOMES:
the viral load | 1 month
  the viral load in the blood of the cord of the newborns infected in utero by CMV the compliance at one month the criteria of tolerance

CONTACTS AND LOCATIONS:
Overall Officials: VILLE YVES, MD, Principal Investigator — Hospital Necker Enfants Malades, Paris France
Locations (1):
- Hospital Necker Enfants Malades, Paris, France

REFERENCES:
- [Background] Bourgon N, Fitzgerald W, Aschard H, Magny JF, Guilleminot T, Stirnemann J, Romero R, Ville Y, Margolis L, Leruez-Ville M. Cytokine Profiling of Amniotic Fluid from Congenital Cytomegalovirus Infection. Viruses. 2022 Sep 28;14(10):2145. doi: 10.3390/v14102145. PMID 36298700
- [Background] Leruez-Ville M, Ghout I, Bussieres L, Stirnemann J, Magny JF, Couderc S, Salomon LJ, Guilleminot T, Aegerter P, Benoist G, Winer N, Picone O, Jacquemard F, Ville Y. In utero treatment of congenital cytomegalovirus infection with valacyclovir in a multicenter, open-label, phase II study. Am J Obstet Gynecol. 2016 Oct;215(4):462.e1-462.e10. doi: 10.1016/j.ajog.2016.04.003. Epub 2016 Apr 13. PMID 27083761
- [Derived] Faure-Bardon V, Magny JF, Parodi M, Couderc S, Garcia P, Maillotte AM, Benard M, Pinquier D, Astruc D, Patural H, Pladys P, Parat S, Guillois B, Garenne A, Bussieres L, Guilleminot T, Stirnemann J, Ghout I, Ville Y, Leruez-Ville M. Sequelae of Congenital Cytomegalovirus Following Maternal Primary Infections Are Limited to Those Acquired in the First Trimester of Pregnancy. Clin Infect Dis. 2019 Oct 15;69(9):1526-1532. doi: 10.1093/cid/ciy1128. PMID 30596974